CLINICAL TRIAL: NCT06924216
Title: Clinical and Radiographic Evaluation of Using Iliac Crest Graft With and Without Platelet-Rich Fibrin (PRF) in Repair of Congenital Alveolar Cleft
Brief Title: Evaluation of Using Iliac Crest With and Without Platelet-Rich Fibrin in Repair of Congenital Alveolar Cleft
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024/801
Record Dates: First submitted 2025-03-12; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Alveolar Clefts; Alveolar Bone Grafting; Alveolar Bone Loss
Keywords: alveolar clefts; iliac crest; graft; PRF
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Alveolar Bone Grafting

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- with platelet-rich fibrin (Experimental): study group: the patients will be treated with iliac crest bone graft with platelet-rich fibrin
  Interventions: Procedure: alveolar bone grafting Plus Platelet rich fibrin
- without Platelet-rich fibrin (Active Comparator): control group : the patients will be treated with iliac crest bone graft only
  Interventions: Procedure: alveolar bone grafting

INTERVENTIONS:
Procedure: alveolar bone grafting — cancellous iliac crest bone will be harvested following the usual surgical procedure. For patients of group a-PRF, it was mixed with 1 cc of the supernatant previously collected, in order to obtain a cohesive bone graft, easier to manipulate.
  The oral mucosal lining will be closed, and a membrane of PRF (PRF group) will be put over the suture line. The alveolar cleft will be then filled with cancellous iliac crest bone along its entire height. A new membrane of PRF will be placed over the bone graft, in order to enclose and protect it. Finally, muco-periosteal flaps will be advanced and sutured without tension over the alveolar crest
  Other Names: Repair of alveolar clefts
  Arms: without Platelet-rich fibrin
Procedure: alveolar bone grafting Plus Platelet rich fibrin — the PRF group: centrifugation at 1300 rpm during 5 minutes, collection of 1 cc of the supernatant, and centrifugation at 1300 rpm during 3 minutes. Careful removal of the clot and separation from the red blood cell fraction with scissors.
  the Platelet-rich fibrin will be added to the surgical site mixed with the iliac crest bone graft and it will also be used as a membrane before closure of the mucoperiosteal flap
  Other Names: PRF
  Arms: with platelet-rich fibrin

SUMMARY:
A randomized clinical trial aims to evaluate the clinical and radiographic outcomes of the repair of congenital alveolar clefts using Iliac crest graft with and without mixing with platelet-rich fibrin

DETAILED DESCRIPTION:
Alveolar clefts occur in response to deviations from normal development in the growth, exposure, and fusion of the frontal eminence. The most common alveolar portion of the cleft is located between the central incisors and canines. The treatment of alveolar clefts is multidisciplinary and aimed at restoring normal ridge contour and functionality. Surgical wound closure is insufficient to repair bony defects, Additional materials are needed for these types of defects, such as bone grafts. Aim: The aim of this study is to evaluate the efficiency of using iliac crest bone graft with and without platelet-rich fibrin in repair of alveolar clefts. Methodology: This study will be conducted on 16 patients with alveolar clefts. The patients will be divided equally and randomly into 2 groups: Group 1 : 8 patients will be treated with iliac crest bone graft only (control group).Group 2: 8 patients will be treated with iliac crest bone graft with platelet-rich fibrin (study group).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with congenital alveolar cleft who need secondary alveolar cleft repair.
2. Patients who are medically fit for surgery under general anaesthesia

Exclusion Criteria:

1. ASA 4 OR ASA 5 patients
2. Uncooperative patients

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-04-27 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in bucco-lingual thickness of the bone at the recipient site | 3 months and 6 months postoperatively
  Post-operative cone beam computed tomographic radiographs will be done using the Scanora 3DX imaging system using a CMOS flat panel detector with isotropic voxel size 133 µm. The x-ray tube that is used to scan the patients possesses a current intensity of 10 mA, 90 KVp, and a focal spot size of 0.5 mm. The scanning time is 14 seconds of pulsed exposure, resulting in an effective exposure time of 3.2 seconds to scan FOV (field of view) of 14 cm height × 16.5 cm width. The raw DICOM data set images will be imported to the On-Demand software (Cybermed, Seoul, Korea) for secondary reconstruction and image analysis.
  CBCT will be performed, and linear measurements will be obtained in axial, sagittal, and coronal cuts to assess the changes in buccolingual thickness of the bone at the recipient site 3 months and 6 months post-operatively.

SECONDARY OUTCOMES:
Calculation of the volume of bone fill in the recipient site | 6 months postoperative
  The volume of remaining alveolar defect around the bone graft at 6 months will be measured and subtracted from the actual alveolar defect volume to calculate the volume of bone fill. The actual volume of alveolar bone graft will be represented as a percentage of bone fill of the alveolar defect volume (Preoperative alveolar Defect Volume minus Postoperative residual defect volume / Preoperative Alveolar defect volume X 100)
wound dehiscence | immediate, 7 days and 14 days postoperative
  Clinical evaluation for wound dehiscence immediate, 7 days, and 14 days postoperatively to detect any complications such as infection, flap dehiscence, or fistula formation. Then the percentage of cases with soft tissue complications will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed S Hamed, professor, Study Director — Suez Canal University; Osama Antar, professor, Study Director — Suez Canal University; Mohamed A Elsholkamy, professor, Study Director — Suez Canal University; Mohamed Nageh, Dr, Study Director — Suez Canal University; Aliaa E Ebrahim, Principal Investigator — Suez Canal University
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bayerlein T, Proff P, Heinrich A, Kaduk W, Hosten N, Gedrange T. Evaluation of bone availability in the cleft area following secondary osteoplasty. J Craniomaxillofac Surg. 2006 Sep;34 Suppl 2:57-61. doi: 10.1016/S1010-5182(06)60013-9. PMID 17071393